CLINICAL TRIAL: NCT00554658
Title: Quetiapine Induced Neuroplasticity in Schizophrenic Patients: A Combined Transcranial Magnetic Stimulation (TMS) and Voxel-based Morphometry (VBM) Study
Brief Title: Quetiapine Induced Neuroplasticity in First-episode Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Goeran Hajak, Prof. Dr. med., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1443L00015
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): Patients will be taken quetiapine for the treatment of first episode schizophrenia.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Quetiapine will be administered open label as clinically required according to current guidelines. Target dose range: 400 - 800 mg quetiapine per day.
  Other Names: Seroquel IR; Seroquel Prolong

SUMMARY:
Aim of the study is to assess the effect of quetiapine treatment in neuroleptic naive, first-episode schizophrenic patients on aspects of functional and structural neuroplasticity assessed by means of transcranial magnetic stimulation and voxel-based morphometry. Main outcome measure is a change in gray matter density under quetiapine treatment from baseline to steady-state-treatment after 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first episode of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) criteria and no history of neuroleptic medication
* Females and/or males aged 18 to 65 years
* Mild to moderate schizophrenia

Exclusion Criteria:

* Neuroleptic treatment prior to study enrollment
* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Any history of neuroleptic treatment
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. angina pectoris, hypertension, congestive heart failure) as judged by the investigator
* Involvement in the planning and conduct of the study
* History of or evidence of significant brain malformation or neoplasm, head injury, cerebral vascular events, neurodegenerative disorder affecting the brain or prior brain surgery
* Concomitant treatment with psychotropic drugs (e.g. antidepressive agents, anticonvulsants, other neuroleptics) except benzodiazepines or hypnotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change of structural neuroplasticity (i.e. change in gray matter density) under treatment with quetiapine assessed by voxel-based morphometry. | 3 weeks

SECONDARY OUTCOMES:
Change of functional neuroplasticity (i.e. cortical excitability) under quetiapine treatment assessed by paired-pulse TMS | 3 weeks
To evaluate the influence of BDNF gene polymorphisms on clinical effects of quetiapine treatment, cortical excitability and brain morphology | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Goeran Hajak, MD, PhD, Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg, Department of Psychiatry, Regensburg, Germany